CLINICAL TRIAL: NCT04486274
Title: Macroscopic on Site Evaluation (MOLSE) vs Standard Specimen Acquisition of Solid Lesions During EUS-FNB: a Randomized Controlled Trial
Brief Title: Macroscopic on Site Evaluation (MOLSE) vs Standard Specimen Acquisition of Solid Lesions During EUS-FNB
Acronym: MOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Istituto Clinico Humanitas Mater Domini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 10-2020
Record Dates: First submitted 2020-07-17; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Endoscopic Ultrasonography With Tissue Acquisition
MeSH Terms: interventions — di-beta-(morpholinoethyl)selenide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non MOSE arm (Experimental): Three needle passes will be performed for each mass
  Interventions: Other: MOSE
- MOSE arm (Experimental): The endoscopist will perform biopsy until a macroscopic visible core (MVC) will be obtained and specimen will be placed in a container (Container A-MOSE). If the needle passes performed are less than 3 (1 or 2 passes) the specimens acquired in the remnant passes to join standard care of 3 passes, according to ESGE guidelines, will be placed in a second container (Container B).
  Interventions: Other: MOSE

INTERVENTIONS:
Other: MOSE — After each pass, the stylet will be introduced into the needle, the material will be released onto a smear slide, and a macroscopic on-site quality evaluation (MOSE) of the specimen will be performed by the endoscopist.

SUMMARY:
Endoscopic ultrasonography (EUS) with tissue acquisition (TA) is nowadays a well-established technique for the sampling of solid lesions pancreatic and non-pancreatic lesions. Actually the standard methods to obtain sampling in gastrointestinal (GI) and non-GI solid masses is the fine needle aspiration (FNA) performed by endoscopic ultrasonography (EUS). Its sensitivity, specificity and diagnostic accuracy for malignant cytology are actually reported of 85-95%, 95%-98% and 78-95% respectively. These data could be affected by the presence of cytopathologist in endoscopy room during the tissue sampling. The rapid on-site evaluation (ROSE) has been advocated to significantly increase EUS-FNA accuracy. To overcome this problem fine needle biopsy (FNB) for TA to obtain histological specimens was proposed. These needles allow as the acquisition of an histological specimen than the cytological one with FNA needles. Recently, the need to obtain a histological, instead of a cytological, specimen during EUS has become more urgent and necessary due to innovative oncological treatment options. An acquired histological specimen could avoid the need of a cytopathologist in the endoscopic room, diminishing costs, procedures time, number of passes and reducing the additional costs of a possible repeated EUS-FNA, in case of an inconclusive diagnosis.

With the advent of FNB, the macroscopic on-site evaluation (MOSE) of the specimen by the endosonographer was proposed, resulting in a comparable alternative to ROSE.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18, both genders.
* Both in-patient and out-patients.
* Presence of a solid lesion. In the presence of a cystic component, the solid part of the lesion should be more 75% of the total.
* FNB performed by a 22G needle Acquire® (Boston Scientific).
* Tissue acquisition with fanning technique.
* Obtained informed consent.

Exclusion Criteria:

* Patients underwent EUS-FNA with or without ROSE
* Patients underwent EUS-FNB plus ROSE.
* Previous biopsy of the lesion with diagnosis of malignancy
* Presence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma.
* Pregnancy or breast-feeding.
* Patients unable to understand and/or read the consent form.
* Inclusion in other study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
To assess the diagnostic accuracy of EUS-FNB with MOSE vs EUS-FNB alone. | 12 Months
  Diagnostic accuracy will be measure

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal Endoscopy Unit, Castellanza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangiavillano B, Crino SF, Facciorusso A, Di Matteo F, Barbera C, Larghi A, Rizzatti G, Carrara S, Spadaccini M, Auriemma F, Fabbri C, Binda C, Coluccio C, Marocchi G, Staiano T, Conti Bellocchi MC, Bernardoni L, Eusebi LH, Cirota GG, De Nucci G, Stigliano S, Manes G, Bonanno G, Ofosu A, Lamonaca L, Paduano D, Spatola F, Repici A. Endoscopic ultrasound-guided fine-needle biopsy with or without macroscopic on-site evaluation: a randomized controlled noninferiority trial. Endoscopy. 2023 Feb;55(2):129-137. doi: 10.1055/a-1915-5263. Epub 2022 Aug 31. PMID 36044915